CLINICAL TRIAL: NCT01435785
Title: Derivation and Prospective Validation of Four Pharmacokinetic-Pharmacodynamic Models of Propofol in Elderly Patients
Brief Title: Performance Evaluation of Four Pharmacokinetic-Pharmacodynamic(PKPD) Models of Propofol in Elderly Patients
Acronym: TCIGeriatric
Status: Completed | Type: Observational
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Pablo O. Sepulveda, MD Professor, Universidad del Desarrollo
Other Study IDs: Propofol TCI in Geriatric
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Propofol Overdose of Undetermined Intent
Keywords: PKPD; Propofol; TCI; Elderly patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood will be centrifugated, the plasma will be frozen and all the samples where analysed wiht HPLC technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the wide use of propofol target-controlled infusion (TCI) in elderly patients, pharmacokinetic (PK) and pharmacodynamic (PD) models performance has not been prospectively assessed in this population. The aims of this study are to derive four PKPD models using previously published PK parameters sets, and to prospectively assess their performance in elderly people. With the obtained data we propose to build a specific PKPD model for this population.

DETAILED DESCRIPTION:
After BIS® and routine monitors were placed, 14 ASA I-II elderly patients (>65 yr) will be anesthetized with plasma TCI of propofol based on Schnider model. After partial recovery from a bolus dose a remifentanil infusion was started and continued throughout surgery. All BIS and TCI data will be continuously record. Arterial blood samples for propofol assays were collected at 1, 2, 3, 5, 10, 20, 40 and 60 min post-induction, and at 0, 1, 3, 5, and 10 min after stopping the infusion. A three compartment effect site model linked to a Sigmoidal Emax PD model, will be used to fit all the data simultaneously in NONMEM. Median performance errors(MDPE), and median absolute performance errors(MDAPE) were calculated to measure bias and accuracy of each model. Comparisons between models will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years, ASA 1,2

Exclusion Criteria:

* Included less than 70% or more than 130% of ideal body weight
* Neurologic disorder
* Use of psychoactive medication, including alcohol intake during the last 48 hours

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients older than 65 years, ASA 1,2 programed for elective sugery
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo O Sepulveda, MD, Principal Investigator — Clinica Alemana Universidad del Desarrollo
Locations (2):
- Chile (2):
  - Clinica Alemana de Santiago, Santiago
  - Clinica Alemana Santiago, Santiago

IPD SHARING:
Plan to Share IPD: Yes
Open TCI proyect